CLINICAL TRIAL: NCT05346965
Title: Musical Training Programme to Enhance Resilience and Self-esteem Among School-aged Children From Low-income Families: A Pilot Randomised Controlled Trial
Brief Title: Musical Training to Enhance Resilience in Children From Low-income Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Alice Ho Miu Ling Nethersole Hospital (Other)
Responsible Party: Principal Investigator, Cheung Tan, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021.590-T
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Resilience

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Musical training programme (Experimental): Participants in the experimental group received a weekly 1-hour musical training lesson for 6 months delivered by professionally qualified musicians. The participants will be assigned a particular musical instrument to learn, and this is based on their interests as well as their capabilities (i.e., fine motor skills), The training will begin at the lowest level (hitting simple notes) and end at the highest level (able to play an entire song).
  Interventions: Behavioral: Musical training
- Wait-list control group (Active Comparator): To ensure equity of access to potentially effective intervention (i.e. musical training programme), participants in the wait-list control group will receive the same musical training programme as participants in the intervention group after the completion of all assessments.
  Interventions: Behavioral: Musical training

INTERVENTIONS:
Behavioral: Musical training — The musical training intervention comprised songs, rhythm and visual creativity to encourage the children to experience music-making as fun.

SUMMARY:
Child poverty is a prominent global health issue owing to its detrimental impact on a child's physical and psychosocial well-being. Nearly 356 million children lived in extreme poverty globally before the pandemic and this is estimated to worsen significantly. children growing up in poverty are more vulnerable to its effect and have an increased risk of psychosocial and developmental problems than children from affluent families. The impact of poverty is not only immediate during childhood but can persist into adulthood. Previous studies have shown that Chinese children from low-income families reported significantly higher levels of depressive symptoms, lower levels of self-esteem, quality of life, and life satisfaction than children from affluent families.

Recent studies have revealed the promising effects of musical training to promote psychological well-being among children and adolescents and paediatric brain tumour survivors, improving psychosocial skills of children with autism, to enhance the quality of life and psychological health by promoting positive emotions and cognitive and social development.

Promoting the psychological health of school-aged children from low-income families through enhancing their resilience has received limited research attention. Additionally, there is a lack of intervention studies to promote resilience in school-aged children from low-income families. This proposed research, therefore, aims to conduct a pilot randomised controlled trial to determine the feasibility, acceptability and preliminary effects of a musical training programme in enhancing resilience and self-esteem, reducing depressive symptoms and improving the quality of life among children from low-income families.

The findings from the study could inform the policymakers and healthcare professionals in health services design and the importance of advocating the psychological needs of children from low-income families by providing adequate community resources and support. If the programme demonstrates its effectiveness in promoting resilience and self-esteem among children from low-income families, further implementation could be done to maintain its sustainability in the community. Most importantly, the programme may potentially enhance the resilience of the vulnerable children from low-income families to combat poverty and hence break the intergenerational transmission of poverty.

ELIGIBILITY:
Inclusion Criteria:

* Chinese children aged between 8-12 years
* able to read Chinese and communicate in Cantonese
* from low-income families, that is, less than half the median monthly household income or recipients of Comprehensive Social Security Assistance

Exclusion Criteria:

* children who are currently receiving or had received musical training before the study
* children have chronic diseases, cognitive and learning difficulties

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Resilience - Resilience Scale for Children | 6-month follow-up
  Children's resilience will be measured by the Resilience Scale for Children- 10 (RS10) which was developed based on the Resilience Scale originally developed by Wagnild and Young. Total scores ranging from 10 to 40, with higher scores indicate higher levels of resilience.

SECONDARY OUTCOMES:
Level of self-esteem - Rosenberg self-esteem scale | Baseline, and 6-month follow-up
  Levels of self-esteem will be measured by the Chinese version of the Rosenberg self-esteem scale (RSES), which is a tool designed to measure the global self-esteem of children and adolescents. Total scores ranging from 10 to 40, with higher scores indicate higher levels of self-esteem.
Depressive symptoms - Center for Epidemiological Studies Depression Scale | Baseline, and 6-month follow-up
  The Chinese version of the Center for Epidemiological Studies Depression Scale for Children (CES-DC) will be used to assess the participants' depressive symptoms. Total scores ranging from 0 to 60, with higher scores indicate higher level of depressive symptoms.
Quality of life - Pediatric Quality of Life Inventory 4.0 Generic Core | Baseline, and 6-month follow-up
  The Chinese version of the Pediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0) will be used to assess children's quality of life. Total scores ranging from 0 to 100, with higher scores represent better quality of life.
Acceptability and satisfaction | 6-month follow-up
  Acceptability and satisfaction will be determined upon the completion of the intervention using a short one-to-one semi-structured interview, which aims to explore the perception of the children and their parents towards the musical training programme; both children and parents will be asked to comment on their experience and feelings of the program; and to provide recommendation for improvement of the programme.

CONTACTS AND LOCATIONS:
Overall Officials: Ankie Tan Cheung, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No